CLINICAL TRIAL: NCT00457977
Title: Pneumococcal Vaccine Response in COPD
Brief Title: Comparing Two Pneumococcal Vaccines in Adults With Chronic Obstructive Pulmonary Disease
Acronym: PNEUMO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 477; U10HL074424 (NIH)
Record Dates: First submitted 2007-04-05; First posted 2007-04-09 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Pneumococcal; Vaccine; Opsonization; Antibodies
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Pneumococcal Vaccines; 23-valent pneumococcal capsular polysaccharide vaccine; Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pneumovax (PPSV23) (Active Comparator): pneumococcal capsular polysaccharide vaccine (PPSV23) (Pneumovax)
  Interventions: Biological: Pneumovax (PPSV23)
- Prevnar (PCV7) (Active Comparator): diphtheria protein-conjugated vaccine (PCV7) (Prevnar) 1.0 mL dose
  Interventions: Biological: Prevnar (PCV7)

INTERVENTIONS:
Biological: Pneumovax (PPSV23) — Injection
  Other Names: 23-valent pneumococcal capsular polysaccharide vaccine; PPSV23; Pneumovax
  Arms: Pneumovax (PPSV23)
Biological: Prevnar (PCV7) — Injection
  Other Names: 7-valent pneumococcal conjugate vaccine; PCV7; Prevnar
  Arms: Prevnar (PCV7)

SUMMARY:
Pneumococcal disease is a serious bacterial infection that can affect different parts of the body, including the lungs. People with chronic illnesses, such as chronic obstructive pulmonary disease (COPD), have a greater risk of developing pneumonia and meningitis as a result of pneumococcal disease. This study will compare the immune response to two types of pneumococcal vaccines in adults with COPD.

DETAILED DESCRIPTION:
Individuals who are infected with the Streptococcus pneumoniae bacteria may develop pneumococcal disease, a serious disease that kills more people in the United States than all other vaccine-preventable diseases combined. Individuals with COPD, characterized by breathing difficulties due to damaged and obstructed lung airways, may have an increased risk of developing serious complications from pneumococcal disease, including pneumonia and meningitis. Currently, there are two types of pneumococcal vaccines available. The pneumococcal capsular polysaccharide (CPS) vaccine, known as Pneumovax, is typically given to adults 65 years of age or older and to any individuals with a serious health condition, including heart disease, lung disease, and diabetes. The diphtheria protein-conjugated vaccine (PCV7), known as Prevnar, is typically given to infants; however, adults who receive this vaccine may also have a favorable response. The purpose of this study is to compare the immune response to the Pneumovax and Prevnar vaccines in adults with COPD.

This study will enroll adults with mild to moderate COPD. Participants will be randomly assigned to receive either the Pneumovax or Prevnar vaccine. This will involve one or two injections. Blood collection will occur during study visits at Months 1, 12, and 24. Study researchers will contact participants by telephone at Months 6 and 18 to document any pneumococcal infections and any additional pneumococcal vaccinations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD)
* Post-bronchodilator forced expiratory volume at one second

  /forced vital capacity (FEV1/FVC) level less than 70%
* Ten or more pack-years of smoking
* Willing to make return visits to the study clinic and accept telephone contact
* Last pneumococcal vaccination occured at least 5 years prior to study entry

Exclusion Criteria:

* Asthma
* Sensitivity to pneumococcal vaccine
* Known bleeding disorder, or requires long-term anticoagulation therapy
* Presence of chronic disease that may impair pneumococcal vaccine response
* Acute illness requiring antibiotics in the month prior to study entry
* Medical condition that makes survival for 24 months following study entry unlikely
* Pregnant

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2007-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonello Punturieri, MD, Study Director — National Heart, Lung, and Blood Institute (NHLBI)
Locations (18):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Veteran's Administration Medical Center, Birmingham, Alabama
  - LA BioMed at Harbor, University of California, Los Angeles, California
  - University of California San Francisco-Airway Clinical Research Center, San Francisco, California
  - Denver Health Medical Center, Denver, Colorado
  - National Jewish Medical and Research Center, Denver, Colorado
  - Veteran's Administration Medical Center, Denver, Colorado
  - University of Maryland Hospital, Baltimore, Maryland
  - Fallon Clinic, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Veteran's Administration Medical Center, Boston, Massachusetts
  - Veteran's Administration Medical Center, Ann Arbor, Michigan
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Veteran's Administration Medical Center, Minneapolis, Minnesota
  - HealthPartners Research Foundation, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Temple University Lung Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Emphysema Research Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Dransfield MT, Harnden S, Burton RL, Albert RK, Bailey WC, Casaburi R, Connett J, Cooper JA, Criner GJ, Curtis JL, Han MK, Make B, Marchetti N, Martinez FJ, McEvoy C, Nahm MH, Niewoehner DE, Porszasz J, Reilly J, Scanlon PD, Scharf SM, Sciurba FC, Washko GR, Woodruff PG, Lazarus SC; NIH COPD Clinical Research Network. Long-term comparative immunogenicity of protein conjugate and free polysaccharide pneumococcal vaccines in chronic obstructive pulmonary disease. Clin Infect Dis. 2012 Sep;55(5):e35-44. doi: 10.1093/cid/cis513. Epub 2012 May 31. PMID 22652582
- [Derived] Dransfield MT, Nahm MH, Han MK, Harnden S, Criner GJ, Martinez FJ, Scanlon PD, Woodruff PG, Washko GR, Connett JE, Anthonisen NR, Bailey WC; COPD Clinical Research Network. Superior immune response to protein-conjugate versus free pneumococcal polysaccharide vaccine in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2009 Sep 15;180(6):499-505. doi: 10.1164/rccm.200903-0488OC. Epub 2009 Jun 25. PMID 19556517
- See also: Click here for the National Institutes of Health Web site. — http://www.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant's were recruited from 10 medical centers across the US from April 9, 2007 to May 7, 2009.
Period: Overall Study
Arm/Group | Pneumovax (PPSV23) | Prevnar (PCV7)
Started | 90 | 91
1-Month | 88 | 87
1-Year | 69 | 76
2-Year | 62 | 66
Completed | 62 | 66
Not Completed | 28 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pneumovax (PPSV23) | Prevnar (PCV7) | Total
Number analyzed (Participants) | 90 | 91 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (10) | 63 (9) | 64 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 32 | 70
  Male | 52 | 59 | 111
Region of Enrollment [Number; unit: participants]
  United States | 90 | 91 | 181
Forced expiratory volume at one second (FEV1) [Mean (Standard Deviation); unit: LIters (L)] | 1.27 (0.50) | 1.33 (0.53) | 1.30 (0.51)
FEV1 (% Predicted) [Mean (Standard Deviation); unit: percent predicted] | 44.8 (15.1) | 44.9 (14.7) | 44.8 (14.9)
forced expiratory volume at one second/forced vital capacity (FEV1/FVC) [Mean (Standard Deviation); unit: percentage of FEV1/FVC] | 45.0 (12.5) | 45.8 (12.6) | 45.4 (12.5)
Race [Number; unit: participants]
  Caucasian | 68 | 70 | 138
  African American | 18 | 18 | 36
  Asian | 0 | 2 | 2
  Native American | 0 | 1 | 1
  Pacific Islander | 1 | 0 | 1
  More than one | 3 | 0 | 3
Oxygen use at baseline [Number; unit: participants]
  Oxygen User | 29 | 21 | 50
  Non-oxygen user | 61 | 70 | 131
Pack years smoking [Mean (Standard Deviation); unit: pack years] | 54.9 (27.1) | 52.0 (27.6) | 53.4 (27.3)
Current Smoker [Number; unit: participants]
  Current Smoker | 32 | 33 | 65
  Non-Current Smoker | 58 | 58 | 116
Vaccine Naive [Number; unit: participants]
  Vaccine Naive | 42 | 45 | 87
  Previously Vaccinated | 48 | 46 | 94

OUTCOME MEASURES:

1. Primary Outcome: Serotype Opsonization Titers
Description: Opsonophagocytosis activity (OPK) serotype specific geometric means
Time Frame: Measured at Baseline, Months 1, 12, and 24
Population: All participants with blood samples were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Pneumovax (PPSV23) | Prevnar (PCV7)
Number analyzed (Participants) | 90 | 91
titers
  Serotype 4 Baseline | 10.85 [7.46 to 15.79] | 12.63 [8.15 to 19.58]
  Serotype 4 1-Month | 132.51 [79.78 to 220.09] | 908.23 [609.84 to 1352.63]
  Serotype 4 1-Year | 61.79 [35.58 to 107.34] | 268.52 [157.82 to 456.86]
  Serotype 4 2-Year | 69.12 [38.15 to 125.23] | 236.89 [134.53 to 417.13]
  Serotype 6B Baseline | 33.26 [20.7 to 53.45] | 49.76 [31.4 to 78.76]
  Serotype 6B 1-Month | 388.08 [231.39 to 650.89] | 1003.30 [653.40 to 1540.56]
  Serotype 6B 1-Year | 293.06 [129.54 to 405.80] | 476.15 [293.06 to 773.64]
  Serotype 6B 2-Year | 240.32 [126.30 to 457.28] | 322.98 [184.43 to 565.62]
  Serotype 9V Baseline | 37.17 [22.25 to 62.08] | 31.44 [19.72 to 50.14]
  Serotype 9V 1-Month | 267.34 [165.45 to 431.96] | 734.52 [488.94 to 1103.43]
  Serotype 9V 1-Year | 142.22 [81.86 to 247.10] | 443.55 [283.80 to 693.21]
  Serotype 9V 2-Year | 219.35 [122.65 to 392.28] | 432.85 [258.03 to 726.13]
  Serotype 14 Baseline | 138.61 [76.62 to 250.75] | 116.90 [63.07 to 216.69]
  Serotype 14 1-Month | 1895.17 [1207.15 to 2975.32] | 2584.06 [1728.32 to 3863.50]
  Serotype 14 1-Year | 839.72 [493.8 to 1427.96] | 1801.11 [1158.45 to 2800.29]
  Serotype 14 2-Year | 594.09 [357.99 to 985.91] | 1255.24 [786.00 to 2004.63]
  Serotype 18C Baseline | 42.32 [25.25 to 70.93] | 42.81 [26.18 to 70.02]
  Serotype 18C 1-Month | 544.49 [334.23 to 887.02] | 1815.99 [1217.04 to 2709.74]
  Serotype 18C 1-Year | 284.41 [170.67 to 473.97] | 665.09 [447.27 to 988.97]
  Serotype 18C 2-Year | 267.94 [151.74 to 473.14] | 540.01 [361.42 to 806.84]
  Serotype 19F Baseline | 13.71 [8.40 to 22.38] | 16.86 [10.31 to 27.57]
  Serotype 19F 1-Month | 266.49 [155.07 to 457.97] | 193.62 [110.85 to 338.22]
  Serotype 19F 1-year | 116.35 [65.51 to 206.66] | 85.87 [47.26 to 156.03]
  Serotype 19F 2-Year | 134.21 [77.52 to 232.36] | 116.40 [64.04 to 211.57]
  Serotype 23F Baseline | 11.79 [7.59 to 18.33] | 18.35 [11.34 to 29.68]
  Serotype 23F 1-Month | 114.86 [64.88 to 203.35] | 1170.32 [700.32 to 1955.75]
  Serotype 23F 1-Year | 47.75 [26.09 to 87.38] | 407.11 [238.14 to 695.95]
  Serotype 23F 2-Year | 39.97 [22.63 to 70.60] | 266.16 [140.25 to 505.09]

2. Secondary Outcome: Serotype-specific Immunoglobulin G (IgG) Antibody Levels
Description: Serotype-specific immunoglobulin G Geometric Mean IgG antibody levels (ug/ml)
Time Frame: Measured at Baseline, Months 1, 12, and 24
Population: All participants with blood samples were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: ug/ml
Arm/Group | Pneumovax (PPSV23) | Prevnar (PCV7)
Number analyzed (Participants) | 90 | 91
ug/ml
  Serotype 4 Baseline | 0.30 [0.23 to 0.38] | 0.28 [0.21 to 0.37]
  Serotype 4 1-Month | 0.74 [0.54 to 1.01] | 1.95 [1.39 to 2.73]
  Serotype 4 1-Year | 0.43 [0.31 to 0.60] | 0.70 [0.50 to 0.97]
  Serotype 4 2-Year | 0.45 [0.32 to 0.65] | 0.53 [0.38 to 0.75]
  Serotype 6B Baseline | 0.89 [0.73 to 1.09] | 0.90 [0.72 to 1.13]
  Serotype 6B 1-Month | 2.26 [1.65 to 3.09] | 3.19 [2.35 to 4.34]
  Serotype 6B 1-Year | 1.32 [1.02 to 1.72] | 1.77 [1.29 to 2.42]
  Serotype 6B 2-Year | 1.27 [0.95 to 1.69] | 1.33 [0.95 to 1.85]
  Serotype 9V Baseline | 0.83 [0.64 to 1.07] | 0.78 [0.60 to 1.01]
  Serotype 9V 1-Month | 2.72 [1.98 to 3.72] | 4.87 [3.64 to 6.50]
  Serotype 9V 1-Year | 1.53 [1.11 to 2.09] | 2.15 [1.59 to 2.91]
  Serotype 9V 2-Year | 1.37 [0.98 to 1.90] | 1.65 [1.22 to 2.24]
  Serotype 14 Baseline | 2.59 [1.87 to 3.57] | 2.53 [1.77 to 3.61]
  Serotype 14 1-Month | 10.80 [7.47 to 15.61] | 15.73 [11.25 to 22.00]
  Serotype 14 1-Year | 5.76 [3.97 to 8.35] | 7.47 [5.15 to 10.84]
  Serotype 14 2-Year | 4.82 [3.38 to 6.88] | 5.68 [3.75 to 8.58]
  Serotype 18C Baseline | 1.16 [0.88 to 1.53] | 1.07 [0.78 to 1.46]
  Serotype 18C 1-Month | 4.25 [3.11 to 5.82] | 9.65 [7.22 to 12.89]
  Serotype 18C 1-Year | 2.25 [1.59 to 3.19] | 3.74 [2.78 to 5.03]
  Serotype 18C 2-Year | 1.94 [1.38 to 2.72] | 2.77 [2.05 to 3.74]
  Serotype 19F Baseline | 3.20 [2.62 to 3.91] | 3.01 [2.45 to 3.70]
  Serotype 19F 1-Month | 6.79 [5.27 to 8.76] | 7.54 [5.76 to 9.85]
  Serotype 19F 1-year | 4.25 [3.26 to 5.53] | 4.32 [3.37 to 5.52]
  Serotype 19F 2-Year | 3.85 [2.90 to 5.11] | 3.68 [2.74 to 4.94]
  Serotype 23F Baseline | 0.58 [0.45 to 0.75] | 0.74 [0.56 to 0.98]
  Serotype 23F 1-Month | 1.88 [1.29 to 2.73] | 7.76 [5.49 to 10.97]
  Serotype 23F 1-Year | 1.12 [0.80 to 1.55] | 2.73 [1.94 to 3.84]
  Serotype 23F 2-Year | 1.00 [0.72 to 1.39] | 1.99 [1.38 to 2.86]

ADVERSE EVENTS:
Time Frame: 2 Years
Arm/Group | Pneumovax (PPSV23) | Prevnar (PCV7)
Serious Adverse Events (participants affected / at risk) | 27/90 | 32/91
Other Adverse Events (participants affected / at risk) | 58/90 | 54/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pneumovax (PPSV23) (N=90) | Prevnar (PCV7) (N=91)
Intestinal Infectious Disease (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (2)
Viral Infection (Infections and infestations) | 1 (1) | 2 (2)
Oral Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Digestive Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Respiratory Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Benign or Uncertain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Hypercalcemia (Endocrine disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Hypertensive (Vascular disorders) | 0 (0) | 1 (1)
Ischemic Heart Disease (Cardiac disorders) | 1 (1) | 2 (3)
Pulmonary Circulation (Vascular disorders) | 1 (1) | 0 (0)
Other Heart Disease (Cardiac disorders) | 2 (2) | 1 (1)
Atherosclerosis (Vascular disorders) | 1 (2) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 7 (7)
Influenza (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COPD (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 11 (14)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 2 (2) | 1 (2)
Liver Disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Inflammatory diseases of prostate (Renal and urinary disorders) | 1 (2) | 0 (0)
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Skin Infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arthropy (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Osteopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Epistaxis (General disorders) | 0 (0) | 1 (1)
Other Respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Death Unkown Cause (General disorders) | 2 (2) | 3 (3)
Complication from surgery (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple drug intoxication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular Disease (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pneumovax (PPSV23) (N=90) | Prevnar (PCV7) (N=91)
Benign or Uncertain Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (6)
Acute Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 15 (18) | 15 (19)
Skin - Inflammatory (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3)
Arthropathy (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Pain (Nervous system disorders) | 5 (7) | 5 (5)
COPD (Respiratory, thoracic and mediastinal disorders) | 40 (84) | 36 (74)
Rheumatism (Musculoskeletal and connective tissue disorders) | 6 (7) | 7 (11)
Other - Respiratory (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 11 (11)
Sprains (Investigations) | 6 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No